CLINICAL TRIAL: NCT06280131
Title: The Efficacy of Pulse Therapy in Acute Relapse in Multiple Sclerosis Patients: Clinical and Neurophysiology Study.
Brief Title: The Efficacy of Pulse Therapy in Acute Relapse in Multiple Sclerosis Patients:
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Entsar Karem Abd Elazeem, Principal investigator, Assiut University
Other Study IDs: multiple sclerosis and pulse
Record Dates: First submitted 2024-01-09; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; pulse therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This work is aimed to assess the short term effect of pulse therapy on clinical and neurophysiological course before and after pulse therapy in order to understand the possible mechanism of action of steroid therapy on RRMS patients low-dose oral treatment should also be retained for patients in whom this approach seems appropriate

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an inflammatory demyelinating disease of the Central Nervous System (CNS) with a variety of clinical presentations MS affects 2.5 million people worldwide. The profound heterogeneity of MS is not limited to the Symptoms but to neuroradiologic and histologic appearances of lesions and response to therapy.

The terms 'acute attack', 'acute exacerbations', and 'relapses' are used interchangeably and refer to the onset or worsening of neurologic deficits lasting ≥24 hours in the absence of fever or infection. Glucocorticoids are used as first-line treatment for attacks as they provide short-term clinical benefits by reducing the severity and shortening the duration of attacks. Typically, intravenous (IV) methylprednisolone 1 g/day for 3-5 days is given, often followed by an oral course of prednisone beginning at a dose of 60-80 mg/day and then tapered over 2 weeks. Other glucocorticoid considerations are dexamethasone1 and high-dose oral prednisone which appear to be equally effective.

Studies using transcranial magnetic stimulation (TMS) have repeatedly reported white-matter involvement in patients with MS as documented by the prolonged central motor conduction time (CMCT), which can differentiate patients with secondary progressive MS (SPMS) from those with relapsing-remitting MS (RRMS), but didn't correlate with severity or degree of improved motor function after corticosteroid therapy. Also, paired-pulse TMS, when delivered at short interstimulus intervals (ISI) (3-5 ms), the conditioned motor evoked potential (MEP) decreases in amplitude (intracortical inhibition, ICI); besides rMT, AMT, Transcallosal inhibition (TCI)and cortical silent period (CSP).

Previously, electrophysiological and clinical evaluations were performed at the onset of therapy and after the end of treatment using an arbitrary evoked potentials score that found evoked potentials may be useful for monitoring acute Multiple Sclerosis bouts and evaluating the effect of therapy.

However, it is difficult to search for an objective marker of the clinical course, in addition no studies were conducted to evaluate the efficacy and underlying mechanism of pulse therapy on clinical course and outcome of relapsing MS and correlating with these recording changes ( pre and post-pulse therapy) in electrophysiological(both evoked potentials and TMS) studies in relapsing MS. Thus the investigator will conduct this study to understand the mechanism of action of pulse therapy on clinical course and recovery of relapsing MS on short term.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient's clinical history and neuroimaging fulfilling revised McDonald diagnostic criteria of Multiple sclerosis in an acute relapsing episode or attack and could be providing consent for participation in the study, will be included in the study.

Exclusion Criteria:

* -Any patient had an infection or febrile condition.
* Any patient had other co-morbid neurological or psychiatric disorders or systemic disease or had contraindications for receiving pulse therapy (high steroid dose) or showed side effects of steroids or intolerance or seizure.
* Any patient refuses participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any adult patient with clinical history and neuroimaging who is fulfilling revised McDonald diagnostic criteria of Multiple sclerosis in acute relapsing episodes or attacks and could be providing consent for participation in the study, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
to evaluate efficacy of a pulse therapy on clinical outcome | 1 month
  evaluate the efficacy of pulse therapy on pyramidal,sensory,cerebellar,brainstem,sphincter and mental by functional systems score which maximum value 46 point and least value 0

SECONDARY OUTCOMES:
clinical correlation between clinical scales scores and neurophysiological changes(visual evoked potional | after 1 day
  visual evoked potion measured by millisecond,normal value less than 95 millisecond
clinical correlation between clinical scales scores and neurophysiological changes( cortical exitability parameters) | after 1 day
  cortical exitability parameters including resting motor transmision measured by millivolt,active motor transmision measured by millivolt,cortical silent period measured by millisecond and transcallosal inhibition measured millisecond

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol